CLINICAL TRIAL: NCT06511648
Title: A Phase 2, Open-label, Multi-centre, Multi-national Interventional Trial to Evaluate the Efficacy and Safety of Erdafitinib (ERDA) Monotherapy and Erdafitinib (ERDA) and Cetrelimab (CET) Combination as Neoadjuvant Treatment in Cisplatin-ineligible Patients With Muscle-invasive Bladder Cancer (MIBC) Whose Tumours Express Fibroblast Growth Factor Receptor ( FGFR ) Gene Alterations
Brief Title: Erdafitinib Monotherapy or in Combination With Cetrelimab in Muscle-invasive Bladder Cancer Patients With Fibroblast Growth Factor Receptor (FGFR ) Gene Alterations
Acronym: SOGUG-NEOWIN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Oncology Genito-Urinary Group (Other)
Collaborators: Janssen-Cilag Ltd. (Industry); Pivotal S.L. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOGUG-2020-IEC(VEJ)-11; 2022-002586-15 (EudraCT Number); 2024-512573-27-01 (EU CTIS Number)
Record Dates: First submitted 2024-07-15; First posted 2024-07-22 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Muscle-invasive Bladder Cancer
Keywords: Urothelial carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erdafitinib (ERDA) monotherapy (Experimental): Patients will receive treatment neoadjuvant with erdafitinib alone (cohort 1: Erdafitinib) before proceeding to radical cystectomy (RC) (to be performed within 2 - 6 weeks after the end of treatment)
  Interventions: Drug: Erdafitinib monotherapy
- Erdafitinib (ERDA) and Cetrelimab (CET) combination (Experimental): Patients will receive treatment neoadjuvant with erdafitinib + cetrelimab (cohort 2: Erdafitinib + Cetrelimab) before proceeding to radical cystectomy (RC) (to be performed within 2 - 6 weeks after the end of treatment)
  Interventions: Drug: Cetrelimab and Erdafitinib combination

INTERVENTIONS:
Drug: Erdafitinib monotherapy — Patients will receive treatment with erdafitinib alone (cohort 1)
  Arms: Erdafitinib (ERDA) monotherapy
Drug: Cetrelimab and Erdafitinib combination — Patients will receive treatment neoadjuvant with erdafitinib plus cetrelimab intravenously (IV).(cohort 2)
  Arms: Erdafitinib (ERDA) and Cetrelimab (CET) combination

SUMMARY:
Erdafitinib (ERDA) alone or in combination with cetrelimab (CET) as neoadjuvant treatment (prior to surgery) in subjects with muscle-invasive bladder cancer (MIBC) whose tumours express Fibroblast Growth Factor Receptor (FGFR )gene alterations and are ineligible for or refuse cisplatin based neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
The aim of the study is to assess the antitumor activity measured as ypT0 rate, defined as no evidence of residual disease based on pathological review of the surgical specimen (pCR) and tumour downstaging (<ypT2). Patients must have a MIBC (cT2-T4a N0/N1 M0) who harbour selected FGFR alterations stated in the protocol and are either ineligible for or refuse cisplatin-based neoadjuvant chemotherapy, as defined by consensus criteria (see 6.1 Inclusion criteria).

Once it is confirmed that the subjects fulfil the eligibility criteria and have signed the informed consent form, they will receive erdafitinib alone (cohort 1) or erdafitinib in combination with cetrelimab (cohort 2).

Patients will receive neoadjuvant treatment with erdafitinib alone (cohort 1) or erdafitinib plus cetrelimab (cohort 2) before proceeding to Radical Cystectomy (RC) (to be performed within 2 - 6 weeks after the last study drug treatment)

Cohort 1: patients will receive erdafitinib Cohort 2: patients will receive erdafitinib in combination with cetrelimab intravenously (IV)

Radiological assessment: A Computed Tomography /Magnetic Resonance Imaging and/or Positron Emission Tomography (per standard local imaging practices) will be scheduled as follow:

* Basal assessment: during screening period (no more than 28 days before Cycle1, Day 1(C1D1)
* Response assessment: At the end of treatment period allowing time for imaging review in advance of Radical cystectomy (RC).
* Follow-up assessment: an image evaluation must be done at first follow-up visit and thereafter, it will be schedule according to local standards and as clinically indicated.

A local pathological assessment will be done on specimens obtained during RC (for co-primary endpoints). Thereafter, during the follow-up period, pathological assessments will be scheduled according to local standards and as clinically indicated.

Patients with disease progression during the treatment phase will be discontinued from the study and will receive their treatment according to the investigator's judgment and monitored to evaluate Overal Survival .

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent stating that he or she understands the purpose of the study and the procedures involved and agrees to participate in the study.
2. Histologically confirmed diagnosis of MIBC (Stage T2-4a N0/N1 M0) obtained via a diagnostic or maximal Transurethral Resection of Bladder Tumor (TURBT) performed no later than 3 months prior to start the screening visit.
3. Pure or predominant (≥50%) urotelial Cancer (UC) histology as determined at the local site.
4. Age ≥ 18 years.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
6. Decline or ineligible ("unfit") for cisplatin-based chemotherapy
7. Presence of a selected FGFR alteration on analysis of tumour biopsy
8. Adequate organ function
9. No other malignancy
10. Willingness to avoid pregnancy or fathering children

Exclusion Criteria:

1. Clinical evidence of N2-N3 tumours or metastatic bladder cancer.
2. Has tumour with any neuroendocrine or small cell component.
3. Patients who are not considered fit for cystectomy or reject cystectomy.
4. Prior FGFR-targeted or an immune checkpoint inhibitor (antiPD1/PDL1 )systemic therapy.
5. Prior systemic therapy, radiation therapy, or surgery for bladder cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) | After a maximum of 30 weeks from the start of treatment (First Followup visit ) on specimens obtained during radical cystectomy.
  Defined as no evidence of residual disease based on pathological review of the surgical specimen.It is defined as the proportion of patients whose pathological staging was ypT0N0M0 as assessed using specimens obtained post radical cystectomy following the study intervention.
Pathological downstaging response <ypT2 | After a maximum of 30 weeks from the start of treatment (First Followup visit ) on specimens obtained during radical cystectomy.
  Defined as no microscopic evidence of residual disease in the bladder (ypT0) or evidence of non-muscle invasive residual disease including ypTa, ypTis, ypT1, based on histological evaluation of the resected bladder specimen collected during cystectomy (post-treatment)."

SECONDARY OUTCOMES:
Rate of pathological downstaging (pDS) | During treatment (27 months)
  Defined as pathological TNM less than clinical TNM.
Event-free Survival rate. | During follow-up period (36 months)
  Radiographically confirmed disease progression of their cancer, death or any event that prevents the performance of RC, including initiation of any additional therapy prior to RC. Progression will be assessed using computed tomography (CT)/magnetic resonance imaging (MRI) and/or Positron Emission Tomography (PET)-CT (per standard local imaging practices).
Overall Survival | During follow-up period (36 months)
  Defined from the date of study entry until death of any cause.
Overall Response Rate | During treatment (27 months)
  Defined as the percentage of patients with partial or complete response according to Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 criteria.
Adverse events. | During treatment (27 months) and follow-up period (36 months)
  Occurring in the period from the time the patient enters the study (from the signature of consent) until 30 days after the last dose of the investigational treatment erdafitinib and until 100 days after the last dose of the investigational treatment cetrelimab
Rate of delay of surgery | During treatment (27 months) and follow-up period (36 months)
  classed as a delay event if performed > 6 weeks after last dose of treatment

CONTACTS AND LOCATIONS:
Locations (23):
- France (5):
  - CLCC Jean Perrin, Clermont-Ferrand
  - CLCC Léon Bérard, Lyon
  - Institut Mutualiste Montsouris, Paris
  - IUCT, Toulouse
  - Institut Gustave Roussy, Villejuif
- Italy (3):
  - IRCCS San Raffaele Hospital and Scientific Institute, Milan
  - A.O. Ordine Mauriziano, Ospedale Umberto I, Turi
  - Ospedale Molinette, Turin
- Spain (10):
  - Hospital Clínic De Barcelona, Barcelona, Catalonia
  - Hospital De Sabadell (Parc Taulí), Barcelona, Catalonia
  - Complexo Hospitalario Universitario A Coruña, A Coruña, Galicia
  - Hospital Universitario Lucus Augusti, Lugo, Galicia
  - ICO l' Hospitalet, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de Toledo, Toledo
  - Fundación Instituto Valenciano De Oncología, Valencia
  - Hospital Clínico Universitario De Valladolid, Valladolid
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (5):
  - University Hospitals of Morecambe Bay NHS Foundation Trust, Lancaster
  - The Royal Marsden NHS Foundation Trust, London
  - Barts Health NHS Trust, London
  - Charing Cross Hospital, London
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield

IPD SHARING:
Plan to Share IPD: No